CLINICAL TRIAL: NCT02009358
Title: Mental Health Promotion Interventions for Reducing Self-reported Depression and Improving Rates of Early Detection of Depression Among Migrant Workers in China, a Cluster Randomised Controlled Trial
Brief Title: Mental Health Promotion Interventions Among Migrant Workers in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xin Yu, Peking University Institute of Mental Health, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GCY2009
Record Dates: First submitted 2013-12-03; First posted 2013-12-12 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2013-12

CONDITIONS: Depression; Anxiety
Keywords: mental health promotion; depression; migrant workers; China
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mental health promotion group (Experimental)
  Interventions: Other: mental health promotion

INTERVENTIONS:
Other: mental health promotion

SUMMARY:
The goals of this research were to conduct a mental health intervention study for reducing self-reported depression and anxiety among migrant workers in a labor-intensive industry in China and to assess the effectiveness of the integrated mental health interventions aimed at promoting the mental health of migrant workers in labor-intensive industries in China.

ELIGIBILITY:
Inclusion Criteria:

* People who worked in the factory agreed to take participant in this study and could understand the questionnaire.

Exclusion Criteria:

* People who don't want to take participant in the study; People can not understand the questionnaire.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 913 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Reducing rate of self-reported depression in BDI | Change from baseline to one year after

SECONDARY OUTCOMES:
Reducing rate of early detection of depression | change from baseline to one year after

OTHER OUTCOMES:
Reducing rate of self-reported anxiety in BAI | change from baseline to one year after

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yu, Professor, Study Director — +86 13910229255